CLINICAL TRIAL: NCT02372097
Title: A Randomized, Open-label, Crossover Phase 1 Study to Evaluate the Bioequivalence Following a Single Oral Dose Administration of SYR-472 25mg and 50mg Tablets in Healthy Adult Male Subjects
Brief Title: A Phase 1, Bioequivalence Study of SYR-472 25mg and 50mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SYR-472-1005; U1111-1167-0746 (Other: WHO); JapicCTI-152813 (Registry Identifier: JapicCTI); JapicCTI-R160849 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Healthy
MeSH Terms: interventions — trelagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Participants in group A will be orally administered 2 tablets of SYR-472 25 mg in period 1 and 1 tablet of SYR-472 50 mg tablet in period 2, both in a single dose under fasting conditions in the morning.
  Interventions: Drug: SYR-472
- Group B (Experimental): Participants in group B will be orally administered 1 tablet of SYR-472 50 mg in period 1 and 2 tablets of SYR-472 25 mg tablets in period 2, both in a single dose under fasting conditions in the morning.
  Interventions: Drug: SYR-472

INTERVENTIONS:
Drug: SYR-472 — SYR-472 25mg, 50mg

SUMMARY:
The purpose of this study is to investigate the bioequivalence of 2 tablets of SYR-472 25 milligram (mg) and 1 tablet of SYR-472 50 mg administered to healthy adult males.

DETAILED DESCRIPTION:
Bioequivalence of 2 SYR-472 25 mg tablets and 1 SYR-472 50 mg tablet administered to healthy adult males will be investigated in a randomized, open-label, crossover study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who understand the outline of the clinical study and are capable of complying with their responsibilities as participants, as judged by the investigator or sub investigator.
2. Participants who can sign and date the informed consent form before the initiation of the study procedure.
3. Healthy Japanese adult males.
4. Participants who are 20 to 35 years of age at the time of informed consent.
5. Participants who weigh 50.0 kilogram (kg) or more with a body mass index (BMI) of 18.5 to less than 25.0 kilogram per square meter (kg/m^2) in the screening period.

Exclusion Criteria:

1. Participants who were administered any investigational product within 16 weeks (112 days) before the start of the study drug administration in stage 1.
2. Participants who have received SYR-472 in the past.
3. Employees of the study site, their family members, those who are in a dependency relationship with employees of the study site involved in the conduct of the study (for example [e.g.], spouse, parents, children, brothers and sisters), and those who might be coerced to consent to participate in the study.
4. Participants who have poorly controlled, clinically significant abnormalities of the nervous system, cardiovascular system, lung, liver, kidneys, metabolism, gastrointestinal system, urinary system, or endocrinological system, which possibly may affect study participation or study results.
5. Participants who have a positive urine drug test in the screening period.
6. Participants who need to use drugs or foods listed in the table of prohibited concomitant drugs and foods.
7. Participants who have a history of hypersensitivity or allergy to drugs (including SYR-472 and its ingredients).
8. Participants who currently have or recently had (within the past 6 months) gastrointestinal disease that may affect drug absorption (malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [at least once a week] heartburn, surgical intervention [e.g., cholecystectomy]).
9. Participants with a past history of cancer.
10. Participants who are positive for any of the following during the screening period: hepatitis B virus surface antigen (HBsAg), antibody against hepatitis C virus (HCV), human immunodeficiency virus (HIV) antigen, anti-HIV antibody, or serological test for syphilis.
11. Participants with difficulty having blood collected from a peripheral vein.
12. Participants who donated 200 milliliter (mL) or more of whole blood within the 4 weeks (28 days) or 400 mL or more of whole blood within the 12 weeks (84 days) before starting the study drug administration in stage 1.
13. Participants who donated a total of 800 mL or more of whole blood within the 52 weeks (364 days) before starting the study drug administration in stage 1.
14. Participants who donated blood components within the 2 weeks (14 days) before starting the study drug administration in stage 1.
15. Participants who show clinically significant abnormalities in electrocardiogram (ECG) during the screening period or on Day 1 (before the study drug administration).
16. Participants who have laboratory test abnormalities suggestive of a clinically significant primary disease or who have abnormal values in any of the following parameters: alanine aminotransferase (ALT) or aspartate serum transaminase AST exceeding 1.5 times the upper limit of the normal range.
17. Participants who are unlikely to comply with the study protocol or are ineligible for the study for any other reason, as judged by the investigator or sub investigator.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 04 March 2015 to 08 April 2015.
Pre-assignment Details: Healthy male participants were enrolled in 1 of the 2 treatment sequences in either Period 1 or 2: Group A: 25 milligram (mg) tablet in Period 1 followed by 50 mg tablet in Period 2, Group B: 50 mg tablet in Period 1 followed by 25 mg tablet in Period 2.
Groups:
- SYR-472 25 mg + SYR-472 50 mg: SYR-472 25 mg, 2 tablets, orally, on Day 1 of the first intervention period (8 days), followed by at least 13 days washout period, followed by SYR-472 50 mg, tablet, orally on Day 1 of the second intervention period (8 days).
- SYR-472 50 mg + SYR-472 25 mg: SYR-472 50 mg, 1 tablet, orally, on Day 1 of the first intervention period (8 days), followed by at least 13 days washout period, followed by SYR-472 25 mg, 2 tablets, orally on Day 1 of the second intervention period (8 days).
Period: First Intervention Period (8 Days)
Arm/Group | SYR-472 25 mg + SYR-472 50 mg | SYR-472 50 mg + SYR-472 25 mg
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Wash Out Period (13 Days)
Arm/Group | SYR-472 25 mg + SYR-472 50 mg | SYR-472 50 mg + SYR-472 25 mg
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention Period (8 Days)
Arm/Group | SYR-472 25 mg + SYR-472 50 mg | SYR-472 50 mg + SYR-472 25 mg
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The pharmacokinetic (PK) analysis set included all participants who received study drug, satisfied the minimum requirements of the protocol with no significant deviations, and were assessable for PK.
Groups:
- Total: Total of all reporting groups
Arm/Group | SYR-472 25 mg + SYR-472 50 mg | SYR-472 50 mg + SYR-472 25 mg | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.7 (2.64) | 22.3 (3.17) | 23.0 (2.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  Japan | 12 | 12 | 24
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 172.0 (6.93) | 172.8 (7.48) | 172.4 (7.06)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 64.51 (9.707) | 62.79 (6.087) | 63.65 (7.972)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 21.69 (1.866) | 21.05 (1.948) | 21.37 (1.894)
Smoking Classification [Number; unit: participants]
  Never Smoked | 7 | 7 | 14
  Current Smoker | 5 | 4 | 9
  Ex-Smoker | 0 | 1 | 1
Alcohol Classification [Number; unit: participants]
  Drinks a Few Days per Week | 2 | 5 | 7
  Drinks a Few Days per Month | 7 | 4 | 11
  Never Drunk | 3 | 3 | 6
Caffeine Classification [Number; unit: participants]
  Caffeine Consumer | 4 | 2 | 6
  Caffeine Non-Consumer | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-168): Area Under the Plasma Concentration-Time Curve From Time 0 to 168 Hours Postdose for Unchanged SYR-472 (SYR-472Z)
Time Frame: Day 1: pre dose (within 3 hours prior to dosing), and at multiple time points (up to 168 hours) post dose in each period
Population: The PK analysis set included all participants who received study drug, satisfied the minimum requirements of the protocol with no significant deviations, and were assessable for PK.
Measure: Geometric Mean (Standard Deviation); unit: nanogram hour per milliliter(ng*hr/mL)
Groups:
- SYR-472 25 mg: SYR-472 25 mg, 2 tablets, once orally, on Day 1 of either Period 1 or Period 2. A washout of 13 days was maintained between the two periods.
- SYR-472 50 mg: SYR-472 50 mg, tablet, once orally, on Day 1 of either Period 1 or Period 2. A washout of 13 days was maintained between the two periods.
Arm/Group | SYR-472 25 mg | SYR-472 50 mg
Number analyzed (Participants) | 24 | 24
nanogram hour per milliliter(ng*hr/mL) | 2733 (445.48) | 2780 (437.95)
Statistical Analysis 1: Comparison: SYR-472 25 mg vs SYR-472 50 mg; The 2-sided 90% confidence interval for the difference between the products (2 tablets of SYR-472 25 mg, 1 tablet of SYR-472 50 mg) was determined from the ANOVA model with the natural logarithms of the AUC(0-168) as a dependent variable, and product, group and period as fixed effects; Test type: Non-Inferiority or Equivalence — Two tablets of SYR-472 25 mg and 1 tablet of SYR-472 50 mg were considered bioequivalent if 90% CI of the mean differences of natural log-transformed AUC(0-168) of SYR-472Z was within the range of ln(0.80) to ln(1.25) or within the range of ln(0.9) to ln(1.11) and the results of dissolution test satisfied the requirement; Least square (LS) mean difference = -0.0170, 90% CI 2-sided [-0.0344 to 0.0004]

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for SYR-472Z
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter(ng/mL)
Arm/Group | SYR-472 25 mg | SYR-472 50 mg
Number analyzed (Participants) | 24 | 24
nanogram per milliliter(ng/mL) | 196.5 (54.034) | 223.6 (67.200)
Statistical Analysis 1: Comparison: SYR-472 25 mg vs SYR-472 50 mg; The 2-sided 90% confidence interval for the difference between the products (2 tablets of SYR-472 25 mg, 1 tablet of SYR-472 50 mg) was determined from the ANOVA model with the natural logarithms of the Cmax as a dependent variable, and product, group and period as fixed effects; Test type: Non-Inferiority or Equivalence — Two tablets of SYR-472 25 mg and 1 tablet of SYR-472 50 mg were considered bioequivalent if 90% CI of the mean differences of natural log-transformed Cmax of SYR-472Z was within the range of ln(0.80) to ln(1.25) or within the range of ln(0.9) to ln(1.11) and the results of dissolution test satisfied the requirement; LS mean difference = -0.1292, 90% CI 2-sided [-0.2177 to -0.0406]

3. Secondary Outcome: AUC(0-inf): Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for SYR-472Z
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SYR-472 25 mg | SYR-472 50 mg
Number analyzed (Participants) | 24 | 24
ng*hr/mL | 2829 (466.32) | 2889 (454.46)
Statistical Analysis 1: Comparison: SYR-472 25 mg vs SYR-472 50 mg; The 2-sided 90% confidence interval for the difference between the products (2 tablets of SYR-472 25 mg, 1 tablet of SYR-472 50 mg) was determined from the ANOVA model with the natural logarithms of the AUC(0-inf) as a dependent variable, and product, group and period as fixed effects; Test type: Superiority or Other; LS mean difference = -0.0210, 90% CI [-0.0362 to -0.0058]

4. Secondary Outcome: Tmax: Time to Reach the Cmax for SYR-472Z
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour(hr)
Arm/Group | SYR-472 25 mg | SYR-472 50 mg
Number analyzed (Participants) | 24 | 24
hour(hr) | 1.5000 [0.50 to 6.00] | 1.000 [0.50 to 6.00]
Statistical Analysis 1: Comparison: SYR-472 25 mg vs SYR-472 50 mg; The 2-sided 90% confidence interval for the difference between the products (2 tablets of SYR-472 25 mg, 1 tablet of SYR-472 50 mg) was determined from the ANOVA model with Tmax as a dependent variable, and product, group and period as fixed effects; Test type: Superiority or Other; LS mean difference = 0.3750, 90% CI 2-sided [-0.1452 to 0.8952]

5. Secondary Outcome: MRT: Mean Residence Time From Time Zero to Infinity for SYR-472Z
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: hr
Arm/Group | SYR-472 25 mg | SYR-472 50 mg
Number analyzed (Participants) | 24 | 24
hr | 32.52 (4.7575) | 33.07 (4.8613)
Statistical Analysis 1: Comparison: SYR-472 25 mg vs SYR-472 50 mg; The 2-sided 90% confidence interval for the difference between the products (2 tablets of SYR-472 25 mg, 1 tablet of SYR-472 50 mg) was determined from the ANOVA model with the natural logarithms of the MRT as a dependent variable, and product, group and period as fixed effects; Test type: Superiority or Other; LS mean difference = -0.0168, 90% CI 2-sided [-0.0504 to 0.0169]

6. Secondary Outcome: Apparent Terminal Elimination Rate Constant (λz) for SYR-472Z
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: per hour(hr-1)
Arm/Group | SYR-472 25 mg | SYR-472 50 mg
Number analyzed (Participants) | 24 | 24
per hour(hr-1) | 0.01399 (0.0036008) | 0.01254 (0.0028378)
Statistical Analysis 1: Comparison: SYR-472 25 mg vs SYR-472 50 mg; The 2-sided 90% confidence interval for the difference between the products (2 tablets of SYR-472 25 mg, 1 tablet of SYR-472 50 mg) was determined from the ANOVA model with the natural logarithms of the λz as a dependent variable, and product, group and period as fixed effects; Test type: Superiority or Other; LS mean difference = 0.1099, 90% CI 2-sided [0.0235 to 0.1963]

7. Secondary Outcome: Number of Participants Reporting One or More Treatment-Emergent Adverse Events (TEAEs)
Description: Collection of AEs commenced from the time that the participant was first administered study drug in Period 1 (Day 1). Routine collection of AEs continued until the end (hospital discharge) of Period 2 (Day 29).
Time Frame: Day 1 of Period 1 up to the day of hospital discharge (Day 29) in Period 2
Population: The safety analysis set included all participants who received study drug.
Measure: Number; unit: participants
Arm/Group | SYR-472 25 mg | SYR-472 50 mg
Number analyzed (Participants) | 24 | 24
participants | 0 | 0

8. Secondary Outcome: Number of Participants With TEAEs Related to Vital Signs
Time Frame: Day 1 of Period 1 up to the day of hospital discharge (Day 29) in Period 2
Population: The safety analysis set included all participants who received study drug.
Measure: Number; unit: participants
Arm/Group | SYR-472 25 mg | SYR-472 50 mg
Number analyzed (Participants) | 24 | 24
participants | 0 | 0

9. Secondary Outcome: Number of Participants With TEAEs Related to Body Weight
Time Frame: Day 1 of Period 1 up to the day of hospital discharge (Day 29) in Period 2
Population: The safety analysis set included all participants who received study drug.
Measure: Number; unit: participants
Arm/Group | SYR-472 25 mg | SYR-472 50 mg
Number analyzed (Participants) | 24 | 24
participants | 0 | 0

10. Secondary Outcome: Number of Participants With TEAEs Categorized Into Investigations System Organ Class (SOC) Related to Laboratory Values
Time Frame: Day 1 of Period 1 up to the day of hospital discharge (Day 29) in Period 2
Population: The safety analysis set included all participants who received study drug.
Measure: Number; unit: participants
Arm/Group | SYR-472 25 mg | SYR-472 50 mg
Number analyzed (Participants) | 24 | 24
participants | 0 | 0

11. Secondary Outcome: Number of Participants Who Had Abnormal and Clinically Significant 12-lead Electrocardiograms (ECG) Findings After Study Drug Administration
Description: Participants whose results of electrocardiograms were judged as abnormal and clinically significant by investigator after study drug administration were counted in this measure.
Time Frame: Baseline up to 7 days after the last dose of study drug (Day 8) in each period
Population: The safety analysis set included all participants who received study drug.
Measure: Number; unit: participants
Arm/Group | SYR-472 25 mg | SYR-472 50 mg
Number analyzed (Participants) | 24 | 24
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 of Period 1 up to the day of hospital discharge (Day 29) in Period 2
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | SYR-472 25 mg | SYR-472 50 mg
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.